CLINICAL TRIAL: NCT02463578
Title: Immunogenicity of a Combined Anti-pneumococcal Vaccine Schedule in Patients With ANCA-associated Vasculitis: a Pilot Study Following New Vaccine Recommendations. PneumoVas Pilot 2
Brief Title: Immunogenicity of a Combined Anti-pneumococcal Vaccine Schedule in Patients With ANCA-associated Vasculitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI15002
Record Dates: First submitted 2015-05-12; First posted 2015-06-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-12

CONDITIONS: Pneumococcal Infection; ANCA-associated Vasculitis
Keywords: Pneumococcal infection; Invasive pneumococcal disease (IPD); Pneumococcal vaccine; Vaccinology; Immunocompromised; Auto-immune diseases; Systemic vasculitis; ANCA-associated vasculitis
MeSH Terms: conditions — Pneumococcal Infections; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Systemic Vasculitis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Exploratory study of anti-pneumococcal immune response in patients with Anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV) immunized according to new vaccine recommendations (i.e. with a combined vaccine schedule (13-valent conjugate pneumococcal vaccine -PCV13- followed by a 23-valent non-conjugate pneumococcal vaccine -PPV23- 8 weeks later).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether this vaccination schedule induces sufficient protective immunity (serotype-specific enzyme linked immunosorbent assay (ELISA) and opsonophagocytosis (OPA) response rates) in AAV-patients receiving immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ANCA-associated vasculitis: diagnosis of granulomatosis with polyangiitis, microscopic polyangiitis or eosinophilic granulomatosis with polyangiitis according to American College of Rheumatology criteria
* Indication for pneumococcal vaccination according to French recommendations (statement of the Haut Conseil de Santé Publique regarding pneumococcal vaccination for adults and children older than 2 years old at risk for invasive pneumococcal disease, April 25Th 2013)

Exclusion Criteria:

* History of pneumococcal immunization 36 months to 24hours before VO.
* Patients with known, or suspected pregnancy
* Patients planning to get pregnant in the year following inclusion
* Splenectomy
* Eosinophilic granulomatosis with polyangiitis (EGPA, Churg-Strauss) flare
* Infection during the week before inclusion
* Patient without social security coverage
* Individuals opposal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for ANCA-associated Vasculitis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Anti-pneumococcal immunity after combined anti-pneumococcal immunization | visit V1 (12 to 16 weeks after V0 (Day 0))
  Proportion of responder patients at V1 (12-weeks after PCV13 injection) to at least 6 of the 10 shared serotypes (i.e. 3, 4, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) included both in PCV13 and PPV23. A serotype is considered positive if the ELISA immunoglobulins G (IgG) antibody titter shows a two-fold increase from baseline (V0) to V1 and is ≥ 1 μg/ml

SECONDARY OUTCOMES:
To assess serotype 3, 4, 6B, 7F, 9V, 14, 18C, 19 A, 19F and 23F-specific immune responses after vaccination | visit V0 (Day 0), visit V1 (12 to 16 weeks after V0) and visit V2 (48 to 56 weeks after V0).
  ELISA specific antibody titres to serotype 3, 4, 6B, 7F, 9V, 14, 18C, 19 A, 19F and 23F.
To assess serotype coverage increase after PPV23 injection | visit V0 (Day 0), visit V1 (12 to 16 weeks after V0) and visit V2 (48 to 56 weeks after V0).
  Serotype 10A and 12F (e.g. 2 PPV23-specific serotypes) ELISA antibody concentrations
For the following serotypes (4, 6B, 9V, 14, 18C, 19F and 23F), to assess the proportion of ELISA-responding patients who also show in vitro opsonophagocytic antibody activity. | visit V0 (Day 0), visit V1(12 to 16 weeks after V0) and visit V2 (48 to 56 weeks after V0).
  For each of the following serotypes (4, 6B, 9V, 14, 18C, 19F and 23F), OPA titers will be measured in ELISA-responding patients at V0, V1, V2. Opsonophagocytic antibody activity is considered positive if the antibody titer shows a four-fold increase from V0 and is above a serotype-specific predefined threshold.
Change Outcome Measures-To assess the sustainability and evolution over time of the vaccine-induced immune response (ELISA and OPA) | visit V2 (48 to 56 weeks after V0).
  For ELISA-responding patients at V1, antibody ELISA concentrations and OPA titers will be measured 52 weeks after PCV13 injection (V2).
Composite Outcome Measures - To identify epidemiologic, clinic and biologic predictive factors that may influence vaccine-induced immune response. | visit V0 (Day 0), visit V1 (12 to 16 weeks after V0) and visit V2 (48 to 56 weeks after V0).
  Analysis of epidemiological, clinical and biological data collected during follow-up: age, sex, history of immunosuppressive therapy, time since previous PPV23 injection, number of previous PPV23 immunizations, AAV activity and severity according to Birmingham Vasculitis Activity Score and Vasculitis Damage Index, results of biological analyses

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Groh, MD, MSc, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP ; Cochin Hospital, Paris, Île-de-France Region, France